CLINICAL TRIAL: NCT01859013
Title: BMI Reduction With Meal Replacements + Topiramate in Adolescents With Severe Obesity
Brief Title: Topiramate in Adolescents With Severe Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1304M31241
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Obesity, Morbid; Obesity; Weight Loss
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss | interventions — Topiramate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Four (4) weeks of meal replacement therapy, followed by 28-weeks of topiramate therapy. Topiramate will be initiated at a dose of 25 mg (taken orally once daily in the evening), escalated to 50 mg (taken orally once daily in the evening) after 1 week, and escalated to 75 mg (taken orally 25 mg in the morning and 50 mg in the evening) after 2 weeks.
  Interventions: Drug: Topiramate
- Sugar Pill (Placebo Comparator): Four (4) weeks of meal replacement therapy, followed by 28-weeks of placebo (sugar pill) therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate will be initiated at a dose of 25 mg (taken orally once daily in the evening), escalated to 50 mg (taken orally once daily in the evening) after 1 week, and escalated to 75 mg (taken orally 25 mg in the morning and 50 mg in the evening) after 2 weeks. Patients who do not tolerate dose escalation will be reduced to the highest tolerated dose for the remainder of the trial.
  Other Names: Topamax
  Arms: Topiramate
Other: Placebo — Placebo will be taken orally once daily in the evening for the first two weeks, and orally twice daily (AM and PM) for the remainder of the study.
  Other Names: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
The prevalence of severe pediatric obesity is on the rise and youth with this condition are at elevated risk for developing chronic diseases such as cardiovascular disease (CVD) and type 2 diabetes mellitus (T2DM). Topiramate, a medication approved by the Food and Drug Administration (FDA) for the treatment of seizures in adults and children, is associated with weight loss. Although not FDA approved for the treatment of obesity, studies in obese adults have demonstrated weight reduction of approximately 5% with 6-12 months of therapy. However, the weight loss effect of topiramate has never been evaluated among children and adolescents. Therefore, the goal of this pilot study is to evaluate the safety and efficacy of 24 weeks of topiramate therapy with a 4-week run-in of meal replacement therapy in adolescents with severe obesity. The primary hypothesis is that 4 weeks of meal replacement therapy followed by 24 weeks of topiramate will have a larger average percent decline in BMI between baseline and 28 weeks compared to meal replacement therapy followed by placebo.

DETAILED DESCRIPTION:
The prevalence of severe pediatric obesity is on the rise and youth with this condition are at elevated risk for developing chronic diseases such as cardiovascular disease (CVD) and type 2 diabetes mellitus (T2DM). Lifestyle modification therapy alone is ineffective for most adolescents with severe obesity and few patients qualify for bariatric surgery. Many patients would likely benefit from pharmacotherapy but only one medication (orlistat) is approved for use in adolescents but notable side effects and limited efficacy impede its clinical use. Topiramate, a medication approved by the Food and Drug Administration (FDA) for the treatment of seizures in adults and children, is associated with weight loss. Although not FDA approved for the treatment of obesity, studies in obese adults have demonstrated weight reduction of approximately 5% with 6-12 months of therapy. However, the weight loss effect of topiramate has never been evaluated among children and adolescents. Therefore, the goal of this pilot study is to evaluate the safety and efficacy of 24 weeks of topiramate therapy with a 4-week run-in of meal replacement therapy in adolescents with severe obesity.

This will be a 28-week, randomized, double-blind, placebo-controlled, pilot clinical trial of meal replacement therapy (4 weeks) followed by topiramate (24 weeks) vs. meal replacement therapy (4 weeks) followed by placebo (24 weeks) for BMI reduction and cardiometabolic risk factor improvement in 36 adolescents (ages 12-17 years old) with severe obesity. Monthly lifestyle modification/behavioral counseling will be delivered by trained study coordinators to patients in both groups. The lifestyle modification education materials will be given to patients and selected sections will be discussed at each monthly contact (five face-to-face sessions and three phone sessions).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥1.2 times the 95th percentile (based on gender and age) or BMI ≥35 kg/m2
* 12-18 years old
* Tanner stage IV or V by physical exam

Exclusion Criteria:

* Tanner stage I, II, or III
* Type 1 or 2 diabetes mellitus
* Previous (within 6-months) or current use of weight loss medication (patients may undergo washout)
* Previous (within 6-months) or current use of drugs associated with weight gain (e.g. steroids/anti-psychotics)
* Previous bariatric surgery
* Recent initiation (within 3-months) of anti-hypertensive or lipid medication
* Previous (within 6-months) or current use of medication to treat insulin resistance or hyperglycemia (patients may undergo washout)
* Major psychiatric disorder
* Females: Pregnant, planning to become pregnant, or unwilling to use 2 or more acceptable methods of contraception when engaging in sexual activity throughout the study
* Tobacco use
* Liver/renal dysfunction

  * ALT or AST >2.5 times the upper limit of normal
  * Bicarbonate <18 mmol/L
  * Creatinine >1.2 mg/dL
* Glaucoma
* Obesity associated with genetic disorder (monogenetic obesity)
* Hyperthyroidism or uncontrolled hypothyroidism
* History of suicidal thought/attempts
* History of kidney stones
* History of cholelithiasis
* Current use of other carbonic anhydrase inhibitor

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Fox CK, Kaizer AM, Rudser KD, Nathan BM, Gross AC, Sunni M, Jennifer Abuzzahab M, Schwartz BL, Kumar S, Petryk A, Billington CJ, Ryder JR, Kelly AS. Meal replacements followed by topiramate for the treatment of adolescent severe obesity: A pilot randomized controlled trial. Obesity (Silver Spring). 2016 Dec;24(12):2553-2561. doi: 10.1002/oby.21633. Epub 2016 Nov 3. PMID 27807925

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 subjects enrolled and 30 were started on the study medication or placebo
Period: Overall Study
Arm/Group | Topiramate | Sugar Pill
Started | 16 | 14
Completed | 12 | 9
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Sugar Pill | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 14 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.6) | 15.7 (1.8) | 15.2 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Mass Index at 28-Weeks
Description: The Percent Change from Baseline in Body Mass Index at 28-Weeks
Time Frame: Baseline and 28-Weeks
Measure: Mean (Standard Deviation); unit: % change BMI
Arm/Group | Topiramate | Sugar Pill
Number analyzed (Participants) | 16 | 14
% change BMI | -2.74 (3.74) | -0.85 (5.31)

ADVERSE EVENTS:
Arm/Group | Topiramate | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes